CLINICAL TRIAL: NCT06598774
Title: Does Smartphone Addiction Affect Cervical Spine Mobility, Head Posture, Body Awareness, and Pain Pressure Threshold?
Brief Title: Cervical Parameters and Body Awareness in Relation to Smartphone Addiction
Status: Completed | Type: Observational
Sponsor: Nagihan Acet (Other)
Responsible Party: Sponsor-Investigator, Nagihan Acet, Asst. Prof., Atılım University
Organization: Atılım University (Other)
Other Study IDs: Atılım Üniversitesi
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Smartphone Addiction
Keywords: Smartphone; Cervical vertebrae; Range of motion; Pain
MeSH Terms: conditions — Internet Addiction Disorder; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Smartphone addiction group: Participants with smartphone addiction
  Interventions: Other: Assessment of head posture:; Other: Assessment of Cervical Pain Pressure Threshold; Other: Assessment of general cervical mobility; Other: Assessment of upper cervical mobility; Other: Assessment of Body Awareness
- Control Group: Participants without smarthone addiction
  Interventions: Other: Assessment of head posture:; Other: Assessment of Cervical Pain Pressure Threshold; Other: Assessment of general cervical mobility; Other: Assessment of upper cervical mobility; Other: Assessment of Body Awareness

INTERVENTIONS:
Other: Assessment of head posture: — Head posture was assessed using photographic methods and craniovertebral angle
Other: Assessment of Cervical Pain Pressure Threshold — The cervical PPTs were assessed using a mechanical pressure algometer (Baseline Force Gauge Model 12-0304; Baseline, NY, USA).
Other: Assessment of general cervical mobility — Cervical mobility was assessed using the CROM (Cervical Range of Motion) deluxe device.
Other: Assessment of upper cervical mobility — It will be assessed using the CROM device and the flexion-rotation test.
Other: Assessment of Body Awareness — Body awareness will be assessed using a questionnaire designed to determine normal or abnormal sensitivity levels in body composition.

SUMMARY:
The study was planned as a observational, cross-sectional study

ELIGIBILITY:
Inclusion Criteria:

* being a smartphone user
* being between the ages of 18 and 25

Exclusion Criteria:

* neck pain
* radicular pain
* neurological symptoms
* cervical surgery or cervical trauma

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consists of smartphone users aged between 18 and 25.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-09-18 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Assessment of Body Awareness | Day 1
  Body awareness will be assessed using a questionnaire designed to determine normal or abnormal sensitivity levels in body composition. The questionnaire consists of four subgroups: 1) Changes in body processes, 2) Sleep-wake cycle, 3) Prediction of disease onset, and 4) Prediction of body responses, with a total of 18 items. Participants were asked to rate each item using a scale from 1 to 7. It has a minimum score of 18 and a maximum score of 126, with higher scores indicating greater body awareness. The validity and reliability of this questionnaire have been reported to be high.
Assessment of head posture | Day 1
  Head posture will be assessed using photographic methods and craniovertebral angle. The craniovertebral angle is calculated as the angle between a horizontal line passing through C7 and a line extending from the tragus of the ear to C7 [23]. An angle less than 49 degrees indicates an anterior head position.
Assessment of Cervical Pain Pressure Threshold (PPT) | Day 1
  The cervical PPTs will be assessed using a mechanical pressure algometer (Baseline Force Gauge Model 12-0304; Baseline, NY, USA). A force will be applied perpendicularly to a 0.5 cm² area at an approximate rate of 3 N/s. While the patient is seated, pressure is applied at the midpoint of the upper trapezius muscle, and 2 cm lateral to the C2 spinous process bilaterally [25]. For each area, two measurements are taken at intervals, and the average of these measurements is calculated to determine the final value.
Assessment of general cervical mobility | Day 1
  Cervical mobility will assessed using the CROM (Cervical Range of Motion) deluxe device, developed by the University of Minnesota. The CROM is an inclinometer system that utilizes gravity and magnetic effects [26]. It is validated for accuracy and reliability. The device consists of two fixed inclinometers for the sagittal and frontal planes, a horizontal inclinometer with a magnetic needle mounted on the top of the device, a magnetic neck brace, a scale-equipped arm with a ruler mounted on the top, and a vertebra locator arm with a weighing system.
Assessment of upper cervical mobility | Day 1
  The CROM device is securely attached to the participant's head while they lay supine on a treatment table. The evaluator asks the participant to relax while the neck is brought to its maximum cervical flexion. In the full flexion position, the head and neck are passively rotated as far as possible within the limits of comfortable pain or physiological stiffness. The procedure is repeated twice on each side with a 30-second rest between tests. The sensitivity of the flexion-rotation test was found to be 91%, its specificity 90%, and its overall diagnostic accuracy 91% . The cervical flexion-rotation test is an important tool in identifying movement impairment at the C1/2 segment and can be used accurately and reliably even by inexperienced examiners.

CONTACTS AND LOCATIONS:
Locations (1):
- Atılım University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sarraf F, Varmazyar S. Comparing the effect of the posture of using smartphones on head and neck angles among college students. Ergonomics. 2022 Dec;65(12):1631-1638. doi: 10.1080/00140139.2022.2047229. Epub 2022 May 4. PMID 35199629
- [Result] Ruivo RM, Pezarat-Correia P, Carita AI. Cervical and shoulder postural assessment of adolescents between 15 and 17 years old and association with upper quadrant pain. Braz J Phys Ther. 2014 Jul-Aug;18(4):364-71. doi: 10.1590/bjpt-rbf.2014.0027. Epub 2014 Jul 18. PMID 25054381
- [Result] Hanten WP, Lucio RM, Russell JL, Brunt D. Assessment of total head excursion and resting head posture. Arch Phys Med Rehabil. 1991 Oct;72(11):877-80. doi: 10.1016/0003-9993(91)90003-2. PMID 1929804
- [Result] Braun BL, Amundson LR. Quantitative assessment of head and shoulder posture. Arch Phys Med Rehabil. 1989 Apr;70(4):322-9. PMID 2930348
- [Result] Niewiadomski C, Bianco RJ, Afquir S, Evin M, Arnoux PJ. Experimental assessment of cervical ranges of motion and compensatory strategies. Chiropr Man Therap. 2019 Jan 22;27:9. doi: 10.1186/s12998-018-0223-x. eCollection 2019. PMID 30680090
- [Result] Mehling WE, Gopisetty V, Daubenmier J, Price CJ, Hecht FM, Stewart A. Body awareness: construct and self-report measures. PLoS One. 2009;4(5):e5614. doi: 10.1371/journal.pone.0005614. Epub 2009 May 19. PMID 19440300
- [Result] Karaca, S., Vücut farkındalığı anketinin Türkçe uyarlaması: geçerlik ve güvenirlik çalışması. Yayınlanmamış yüksek lisans tezi, Muğla Sıtkı Koçman Üniversitesi Sağlık Bilimleri Enstitüsü, Muğla, 2017.
- [Result] Jung SI, Lee NK, Kang KW, Kim K, Lee DY. The effect of smartphone usage time on posture and respiratory function. J Phys Ther Sci. 2016 Jan;28(1):186-9. doi: 10.1589/jpts.28.186. Epub 2016 Jan 30. PMID 26957754
- [Result] AlZarea, B.K. and S.R. Patil, Mobile phone head and neck pain syndrome: proposal of a new entity. Headache, 2015. 251(63): p. 313-317.